CLINICAL TRIAL: NCT01509157
Title: Prevention of Nocturnal Hypoglycemia in Children and Young Adults With Type 1 Diabetes Using a Remote Safety and Control Diabetes Management System
Brief Title: MDRS for Prevention of Nocturnal Hypoglycemia
Acronym: MDRS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: rmc006447ctil
Record Dates: First submitted 2011-12-25; First posted 2012-01-12 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Continuous Glucose Monitoring; Nocturnal Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MDRS system (Experimental): Participants will be using the MDRS system combined with their regular treatment with Continuous Glucose Monitoring during nightime for 2 weeks. The MDRS will allow the supervising personal to get real time remote data of glucose level and to alarm the patients and intervene in cases such as pending hypoglycemia, long standing hyperglycemia or technical faults
  Interventions: Device: MDRS System (Remote & Safety diabetes management system)
- Continuous Glucose Monitoring (Active Comparator): Participants will be using their regular Continuous Glucose Monitoring during nightime for 2 weeks, without using the MDRS remote control system
  Interventions: Procedure: Continuous Glucose Monitoring

INTERVENTIONS:
Device: MDRS System (Remote & Safety diabetes management system) — Participants will be using the MDRS system combined with their regular Continuous Glucose Monitoring during nightime for 2 weeks. The MDRS will allow the supervising personal to get real time remote data of glucose level and to alarm the patients and intervene in cases such as pending hypoglycemia, long standing hyperglycemia or technical faults
  Arms: MDRS system
Procedure: Continuous Glucose Monitoring — Participants will be using their regular Continuous Glucose Monitoring during nightime for 2 weeks, without using the MDRS remote control system
  Arms: Continuous Glucose Monitoring

SUMMARY:
The investigators have developed a unique Remote & Safety diabetes management system (MDRS) that offers real-time remote monitoring and control of glucose levels. The system allows the supervising personal to alarm the patient and intervene in cases such as pending hypoglycemia, long standing hyperglycemia or technical faults.The aim of this feasibility study is to evaluate the efficacy of the MDRS system in preventing nocturnal hypoglycemia in children and young adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed at least 1 year prior to study entry
* Continuous subcutaneous insulin infusion pump for at least 3 month prior to study entry
* Use of continuous glucose measurement device for at least one month prior to study entry
* Age: 4-24 years old
* HbA1c < =8.5%
* No more than one severe hypoglycemia or an episode diabetic ketoacidosis within the year prior to study entry, and none within the month prior to study entry.
* Capable of reading a pump screen in English
* Capable of operating the MDRS software
* A patient older than 18 years- leaving routinely with at least one more adult(age above 18 years) capable of connecting the C&C center and properly reacting to the instructions given by the attending personal.
* A patient younger than 18 years- leaving routinely with at least two adults (age above 18 years) capable of connecting the C&C center and properly reacting to the instructions given by the attending personal.
* All participants must provide an adult independent contact person, leaving near by the participant, capable of connecting the C&C center and properly reacting to the instructions given by the attending personal. This person will be called into action in emergency cases in which the participant or his household members can not be reached.
* Capable of completing the hypoglycemia the relevant surveys
* Able to understand and sign an informed consent forms

Exclusion Criteria:

* Any significant disease or conditions, including psychiatric disorders that in the opinion of the principal investigator are likely to effect subject compliance or the subjects ability to complete the study.
* Patients participating in other device or drug studies
* Known dermal hypersensitivity to trial products or those that contain medical adhesive
* Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication for participation in the study.
* Inability to understand/complete the hypoglycemia fear survey
* Female subject who is pregnant or planning to become pregnant within the planned study duration

Ages: 4 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduction in time spent in hypoglycemia | 4 weeks (end of study period)
Parental fear of hypoglycemia | 4 weeks ( end of study pariod)

SECONDARY OUTCOMES:
Change in Treatment Satisfaction | between week 0 (baseline) and week 4 (end of study period)
  We will measure the change in Treatment Satisfaction using questioner and calculation of the the satisfaction score
Percentage of time spent in the target range | 4 weeks (end of study period)
  Percentage of time spent in the target range, defined as sensor glucose level within 63-140 mg/dl
Percentage of time spent in the tight normal range | 4 weeks (end of study period)
  Percentage of time spent in the tight normal range, defined as sensor glucose level within 80 to 120 mg/dl
Average and median of blood glucose levels | 4 weeks (end of study period)
Percentage of time spent below 63 mg/dl | 4 weeks (end of study period)
Percentage of time spent above 140,180,250 mg/dl | 4 weeks (end of study period)
Glucose variability | 4 weeks (end of study period)
  Glucose variability measured by glucose Standard Deviation and "Kovatchev indexes"
Hypoglycemic events-number and severity of episodes | 4 weeks (end of study period)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Oron T, Farfel A, Muller I, Miller S, Atlas E, Nimri R, Phillip M. A remote monitoring system for artificial pancreas support is safe, reliable, and user friendly. Diabetes Technol Ther. 2014 Nov;16(11):699-705. doi: 10.1089/dia.2014.0090. Epub 2014 Sep 11. PMID 25211216